CLINICAL TRIAL: NCT02822105
Title: Phase 1 Clinical Study To Investigate The Safety And Immunogenicity Of The H3N2 (A/Brisbane/10/2007) M2SR Monovalent Influenza Vaccine
Brief Title: Safety and Immunogenicity Study of H3N2 M2SR Monovalent Influenza Vaccine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FluGen Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H3N2-V001
Record Dates: First submitted 2016-06-27; First posted 2016-07-04 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Flu
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- H3N2 M2SR monovalent influenza vaccine (Experimental): This group will receive a low, medium or high dose of the H3N2 M2SR monovalent influenza vaccine administered intranasally. It will be compared with placebo in a 3:1 ratio.
  Interventions: Biological: the H3N2 M2SR monovalent influenza vaccine
- placebo (Experimental): This group will receive saline administered intranasally.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: the H3N2 M2SR monovalent influenza vaccine — The H3N2 Bris10 M2SR influenza vaccine candidate (Bris10 M2SR) is formulated to contain different levels of an M2-deleted non-replicating influenza virus expressing the HA and NA genes of influenza strain A/Brisbane/10/2007.
  Arms: H3N2 M2SR monovalent influenza vaccine
Other: Placebo — saline
  Arms: placebo

SUMMARY:
The purpose is of this study is to assess the safety and tolerability of three dose levels of H3N2 M2SR influenza vaccine versus placebo delivered intranasally to healthy adult subjects.

DETAILED DESCRIPTION:
Healthy adult subjects will be screened with the objective to randomize 96 subjects with the lowest levels of H3 hemagglutination inhibition (HAI) titers that meet all inclusion/exclusion criteria and have signed an informed consent. Subjects will be rank ordered from low to high based on their HAI titer. Subjects will then be assigned treatment based on a randomization to either active vaccine or placebo. The first two subjects dosed in each dose cohort will serve as sentinels and will receive active IP (not randomized).

Subjects will receive a single dose inoculation of the H3N2 M2SR seasonal monovalent influenza vaccine administered intranasally as a liquid formulation, or placebo (saline). The sentinel subjects will be vaccinated in dose cohort 1 and a safety monitoring committee (SMC) will conduct a review of safety data, tolerability, reactogenicity, and clearance of infectious virus prior to dosing the remaining subjects of the cohort with active or placebo.

After the last subject in the cohort has been followed for at least 7 days the SMC will conduct another review of safety data prior to proceeding to the next higher dose level: Cohort 2. The same processes of sentinel subject dosing and SMC review will be conducted for Cohorts 2 and 3.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals who are in good health at the time of entry into the study as determined by medical history, physical examination, vital signs, and clinical safety laboratory values and clinical judgement of the Principal Investigator (PI)
* The subject signs and dates a written, informed consent form and any required privacy authorization
* Willing to use a reliable form of contraception approved by the Investigator (e.g., intrauterine device [IUD], female condom, diaphragm with spermicide, cervical cap, use of condom by the sexual partner or a sterile sexual partner) for 1 month prior to vaccination and until 28 days following the last visit
* Individuals who are willing and able to communicate with the Investigator and understand the requirements of the study
* Individuals who can comply with trial procedures and are available for the duration of follow-up

Key Exclusion Criteria:

* Any subject with the following screening lab values (per the Food and Drug Association (FDA) Guidance: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials):

  1. Any ≥ Grade 2 abnormality
  2. Clinically significant Grade 1 abnormality as judged by the Principal Investigator or
  3. Clinically non-significant Grade 1 abnormality as judged by the Principal Investigator which, upon repeat testing becomes more abnormal
* History or clinical manifestation of clinically significant health conditions including but not limited to: mental illness, active hematological, renal, hepatic, pulmonary, central nervous, neurological, cardiovascular, endocrine (including diabetes mellitus) or gastrointestinal disorders
* Acute febrile illness within 72 hours prior to vaccination, defined as the presence of a moderate or severe illness with or without fever (as determined by the Investigator through medical history and physical examination), or presence of a fever >38ºC orally.
* Any confirmed or suspected immunosuppressive or immunodeficient state including: asplenia, recurrent severe infections and chronic (more than 14 days) immunosuppressant medication
* Living in the same household with any person with a non-functional or suppressed immune system

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of local and systemic adverse events (AEs) through 28 days vaccination and cumulatively through Day 180 | from baseline through study completion (Day 180)
  Record adverse events

SECONDARY OUTCOMES:
Percentage of subjects demonstrating seroconversion to vaccine hemagglutinin antigen and the magnitude of the immune response | from baseline through study completion (Day 180)
  Test antibodies pre and post vaccination
Length of time that vaccine virus shedding is detected | at 24, 48 and 72 hours post-vaccination and on day 7 post vaccination
  Test nasal swabs for virus

CONTACTS AND LOCATIONS:
Overall Officials: Renee Herber, Study Director — FluGen Inc; Carlos Fierro, MD, Principal Investigator — Johnson County Clin Trials
Locations (1):
- JCCT, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Publications and post to site